CLINICAL TRIAL: NCT07235501
Title: Kinetic Analysis of Immune Cells in Blood and Chronic Graft-Versus-Host Disease-Affected Tissues After Allogeneic Hematopoietic Cell Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 24871; NCI-2025-04424 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24871 (Other: City of Hope Medical Center); P30CA033572 (NIH); R01HL170099 (NIH)
Record Dates: First submitted 2025-11-10; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Graft Versus Host Disease; Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational Cohort 1: Patients undergo blood, saliva/buccal, and stool sample collection for up to 2 years on study. Patients also have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study
- Observational Cohort 2: Patients undergo a one-time blood, saliva/buccal, and stool sample collection and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study evaluates the factors that contribute to chronic graft-versus-host disease, which is a complication that can occur after allogeneic hematopoietic cell transplantation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Characterize immune cells and their subsets in peripheral blood of patients who develop and do not develop chronic graft-versus-host disease (cGVHD).

OUTLINE: This is an observational study. Patients are assigned to 1 of 2 cohorts.

COHORT 1: Patients undergo blood, saliva/buccal, and stool sample collection for up to 2 years on study. Patients also have their medical records reviewed on study.

COHORT 2: Patients undergo a one-time blood, saliva/buccal, and stool sample collection and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* * BOTH COHORTS:

  * Documented written informed consent of the participant and/or parent/guardian.

    * Assent from pediatric participants will be documented per institutional policies and practice.
  * Patients who have received allogeneic hematopoietic cell transplant (HCT) regardless of donor type, condition regimen, or GVHD prophylaxis.
  * Age: ≥ 18 years or ≥ 7 years if 30 kg and above
  * Willingness to:

    * Provide blood sample(s), stool, saliva, and buccal mucosa,
    * If applicable: Permit medical record/ clinical laboratory result review

      * COHORT 1:
  * Patients who have received allogeneic hematopoietic cell transplant (HCT) regardless of donor type, condition regimen, or GVHD prophylaxis.

    * COHORT 2:
  * Patients diagnosed with cGVHD at any time-point after allogeneic HCT regardless of donor type, condition regimen, or GVHD prophylaxis.

Exclusion Criteria:

* * Women of childbearing potential: Pregnant/nursing

  * Individuals with impaired decision-making capacity
  * An employee who is under the direct/ indirect supervision of the PI/ a co-investigator/ the study manager
  * A direct study team member

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have received allogeneic hematopoietic cell transplant.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2026-01-27 (Estimated); Primary Completion 2028-04-11 (Estimated); Study Completion 2028-04-11 (Estimated)

PRIMARY OUTCOMES:
T cell measurements | Up to 2 years - study completion
  Defined as percentage of naïve and memory T cells using high dimensional flow cytometry.
B cell measurements | Up to 2 years - study completion
  Defined as percentage of naïve B, memory B, and plasma cells using high dimensional flow cytometry.
Macrophage measurements | Up to 2 years - study completion
  Defined as percentage of M1, M2, and M0 using high dimensional flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Nakamura, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States